CLINICAL TRIAL: NCT03421665
Title: A Multicenter, Prospective, Post-Market Clinical Follow-Up Evaluation of the Titan 3-D™ Wedge System
Brief Title: Evaluation of the Titan 3-D™ Wedge System
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decided to pursue an alternative study prior to subject enrollment.
Sponsor: Paragon 28 (Industry)
Responsible Party: Sponsor
Other Study IDs: P03-SP-0001
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Flat Foot; Lateral Column Lengthening; Medial Cuneiform Osteotomy
Keywords: titanium wedge; Evans; Cotton
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Titan 3-D Wedge System: Subjects who receive one or more Titan 3D wedge(s).
  Interventions: Device: Titan 3D Wedge System

INTERVENTIONS:
Device: Titan 3D Wedge System — Each subject will undergo an LCL procedure and/or medial cuneiform osteotomy with one or more TITAN 3-D™ Wedges. Ancillary fixation should be used in conjunction with each TITAN 3-D™ Wedge used. This surgical procedure will be performed as standard of care and is not part of the research procedures. Post-operative care and weight-bearing/activity restrictions will be at the discretion of the surgeon as part of their standard of care for the procedure.

SUMMARY:
Evaluate clinical healing and radiographic maintenance of correction following an LCL procedure or medial cuneiform osteotomy (Cotton) at 6 months following the use of the TITAN 3-D™ Wedge. Subjects who receive one or more TITAN 3-D™ Wedges will obtain satisfactory levels of clinical healing and radiographic maintenance of correction at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has foot pain/discomfort on the foot in question.
2. The subject has activity limitations due to the foot in question.
3. The subject agrees to comply with the requirements of the study and complete the study measures.
4. The subject (or representative of the subject in the case of a minor) is willing and able to provide written informed consent.
5. The subject plans on undergoing an LCL procedure and/or medial cuneiform osteotomy with a TITAN 3-D™ Wedge.

Exclusion Criteria:

1. The subject is pregnant.
2. The subject had been previously sensitized to titanium.
3. The subject is scheduled for a same day bilateral LCL procedure or medial cuneiform osteotomy procedure.
4. The subject is not expected to complete the study according to the investigation plan.
5. The subject has been deemed physiologically or psychologically inadequate by the enrolling physician.
6. The subject is: a prisoner, unable to understand what participation in the study entails, mentally incompetent, a known abuser of alcohol and/or drugs or anticipated to be non-compliant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include males and females of all ages. Furthermore, it is likely that the majority of subjects enrolled in this study suffer from a flatfoot deformity; however, this study will not be restricted to only those diagnosed with flatfoot.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-06-15 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Healing | 6 Months
  Evaluate clinical healing following an LCL procedure or medial cuneiform osteotomy (Cotton) at 6 months following the use of the TITAN 3-D™ Wedge. Clinical healing is defined as lack of pain over the osteotomy site.
Radiographic Maintenance of Correction | 6 Months
  Evaluate radiographic maintenance of correction following an LCL procedure or medial cuneiform osteotomy (Cotton) at 6 months following the use of the TITAN 3-D™ Wedge. Radiographic maintenance of correction is defined as the absence of a clinically relevant change in radiographic measures across post-operative time points.

SECONDARY OUTCOMES:
Time to clinical/radiographic healing (union) | 24 Months
  Evaluate time to clinical/radiographic healing (union vs. non-union) after a Titan 3D wedge procedure
Clinical complications | 24 Months
  Complications due to the procedure
Maintenance of implant position | 24 Months
Maintenance of anatomical alignment | 24 Months
Determine bone reaction, if any, to the device such as overgrowth or cystic lesions | 24 Months
Determine rate of removal of the device and subsequent healing | 24 Months
Change in anatomical and radiographic angular/positional alignment before and after an LCL procedure and/or medial cuneiform osteotomy using a TITAN 3-D™ Wedge | 24 Months
Change in VAS Pain Score across multiple time points | Pre-operatively, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Visual Analog Scale (VAS). Line from 0 (no pain) to 10 (worst pain). Patient reported.
Change in AOFAS Ankle-Hindfoot and/or Midfoot Score across multiple time points | Pre-operatively, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot clinical score.
  Pain: 0-40 points Function: 0-50 points Alignment: 0-10 points Total Score (sum): 0-100 points (higher score indicates better outcomes)
  American Orthopaedic Foot and Ankle Society (AOFAS) Midfoot clinical score. Pain: 0-40 points Function: 0-45 points Alignment: 0-15 points Total Score (sum): 0-100 points (higher score indicates better outcomes)
Change in PROMIS Pain Intensity Score across multiple time points | Pre-operatively, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score, Item Bank v1.0, SF 3a.
  Raw Score Range: 3 (no pain) to 15 (very severe pain)
Change in PROMIS Mobility Score across multiple time points | Pre-operatively, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Mobility Score, Item Bank v2.0.
  Raw Score Range: 15 (high level of difficulty) to 120 (no difficulty)
Change in PROMIS Pain Interference Score across multiple time points | Pre-operatively, 2 weeks, 6 weeks, 12 weeks, 6 months, 12 months, 24 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Score, Item Bank v1.0, SF 6a.
  Raw Score Range: 6 (no interference) to 30 (high level of interference)
Compare the outcomes and complication rates of TITAN 3-D™ Wedges with previously published outcomes of historical controls, allograft bone and autograft bone | 24 Months

IPD SHARING:
Plan to Share IPD: No